CLINICAL TRIAL: NCT00507650
Title: Supplement Fluid & Collagen Deposition
Brief Title: Increasing Fluids in Older Adults to Prevent & Treat Pressure Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NR0008241
Record Dates: First submitted 2007-07-24; First posted 2007-07-26 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Pressure Ulcers
Keywords: Pressure ulcers; Geriatrics; Nursing home; Fluid balance; Collagen deposition
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prescribed (Active Comparator): Fluid volume and type prescribed by MD or provider.
  Interventions: Dietary Supplement: Fluid intervention
- Supplemental (Experimental): Fluid volume and type prescribed by physician or provider plus 10 ml/kg X 5 days.
  Interventions: Dietary Supplement: Fluid intervention plus 10 ml/kg/day

INTERVENTIONS:
Dietary Supplement: Fluid intervention — Volume of fluid prescribed by physician or provider/day X 5 days.
  Arms: Prescribed
Dietary Supplement: Fluid intervention plus 10 ml/kg/day — Fluid volume and type prescribed by physician or provider plus 10 ml/kg/day X 5 days.
  Arms: Supplemental

SUMMARY:
The purpose of this study is to determine whether providing extra fluid to nursing home residents will help prevent or heal pressure ulcers. We hypothesize that providing extra fluid to nursing home residents will increase their skin blood flow and oxygen to support healing and maintaining healthy skin. Participants are enrolled who have a pressure ulcer or who are at-risk for an ulcer (determined by looking at risk factors). The study is divided into two 10 day phases. In Phase 1, we examine participant's usual status, including fluid intake and baseline healing potential. In Phase 2, participants are randomly placed in groups to receive either their usually prescribed fluid intake or additional fluid. A study nurse provides the fluid to the residents. We measure their actual intake, their body water, how well their kidneys are working, their potential to heal, and also monitor them for the development of fluid overload. This study is important because it helps us understand the role of a basic nursing intervention in the prevention and treatment of pressure ulcers.

DETAILED DESCRIPTION:
Pressure ulcers are prevalent in nursing homes. They heal slowly, cause pain, impair quality of life, and are expensive to treat. Dehydration is a problem in some nursing home residents and under-perfusion a problem in others. Theoretically, providing supplemental fluid to under-hydrated residents should increase fluid in the various fluid compartments of the body, increase subcutaneous oxygen, support skin integrity, enhance pressure ulcer blood flow and pressure ulcer healing, including collagen production. This proposition has not been examined in nursing home residents with pressure ulcers.

The purpose of this randomized clinical trial (RCT) in which subjects serve as their own control is to determine whether administration of supplemental fluid to nursing home residents with or at risk for pressure ulcers enhances collagen deposition. Specifically, this study will determine whether oral administration of supplemental fluid given daily for five days to persons with or at risk for pressure ulcers enhances collagen deposition, increases total body water, augments subcutaneous tissue oxygen, increases pressure ulcer oxygenation, and is safe.

The sample will be nursing home residents at risk for or with pressure ulcers. After consent, baseline measures of collagen deposition, pressure ulcer oxygen, fluid intake, and body water in the various fluid compartments are measured. Expanded polytetrafluoroethylene (ePTFE) tubes are used to measure collagen deposition. Bioelectrical impedance is used to measure body water. In the treatment phase, subjects are randomized to one of the two supplemental fluid regimes. Supplemental fluid is administered for five days and collagen deposition, subcutaneous tissue oxygen, pressure ulcer oxygen, and body water in the various compartments again measured. Subjects are monitored for fluid overload. Data are analyzed with RMANOVA and logistic regression techniques.

ELIGIBILITY:
Inclusion Criteria:

* Persons age =/> 60 years at risk for pressure ulcers (Braden Scale score <18 or nonblanchable erythema [Stage 1 ulcer]) or with a Stage II-IV pressure ulcer and WBC of at least 2,000/mm3

Exclusion Criteria:

Those:

* Who have or have had heart failure or renal failure/insufficiency
* Who currently smoke
* With acute illness or having experienced it in the last 7 days
* Taking immunosuppressive drugs
* With an implantable defibrillator
* With a glycosylated hemoglobin of >8%
* With a body mass index is <21 kg/m2 or > 30 kg/m2; and
* Being treated for dehydration.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2003-09; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Collagen deposition | 10 days

SECONDARY OUTCOMES:
Total body water | 10 days
Safety - development of heart failure | Study duration

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A. Stotts, RN, EdD, Principal Investigator — University of California, San Francisco